CLINICAL TRIAL: NCT02019472
Title: A Multicenter, Randomized, Double-blind, Parallel Group Study of Sirukumab Monotherapy Compared With HUMIRA® Monotherapy Administered Subcutaneously, in Subjects With Active Rheumatoid Arthritis
Brief Title: A Study Comparing Sirukumab (CNTO 136) Monotherapy With Adalimumab (HUMIRA®) Monotherapy in the Treatment of Active Rheumatoid Arthritis
Acronym: SIRROUND-H
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR103111; CNTO136ARA3005 (Other: Janssen Research & Development, LLC); 2013-001417-32 (EudraCT Number)
Record Dates: First submitted 2013-12-18; First posted 2013-12-24 (Estimated); Results first posted 2017-09-14 (Actual); Last update posted 2017-10-26 (Actual); Status verified 2017-09

CONDITIONS: Arthritis, Rheumatoid
Keywords: Rheumatoid arthritis; CNTO 136; Sirukumab; Adalimumab; HUMIRA®
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adalimumab; sirukumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1 (adalimumab 40 mg) (Experimental): Adalimumab 40 mg SC at Weeks 0, 2, and every 2 weeks through Week 52. At Week 16, subjects who have < 20% improvement from baseline in both swollen and tender joint counts will early escape in a blinded fashion and receive adalimumab 40 mg every week through Week 52.
  Interventions: Biological: adalimumab 40 mg
- Group 2 (sirukumab 100 mg) (Experimental): Sirukumab 100 mg SC at Weeks 0, 2, and every 2 weeks through Week 52. Subjects may meet the early escape criteria at Week 16 (< 20% improvement from baseline in both swollen and tender joint counts) but no sirukumab dose adjustments will made for these subjects. However, these subjects will receive placebo injections every 2 weeks between the sirukumab injections (ie, subjects that early escape will receive a weekly injection of alternating sirukumab and placebo, to preserve the blind).
  Interventions: Biological: sirukumab 100 mg; Drug: Placebo
- Group 3 (sirukumab 50 mg) (Experimental): Sirukumab 50 mg SC at Weeks 0, 4, and every 4 weeks through Week 52. Between sirukumab injections, placebo SC injections will be administered at Weeks 2, 6, and every 4 weeks through Week 50. At Week 16, subjects who have < 20% improvement from baseline in both swollen and tender joint counts will early escape in a blinded fashion and receive sirukumab 100 mg every 2 weeks through Week 52 and placebo injections every 2 weeks between the sirukumab injections (ie, subjects that early escape will receive a weekly injection of alternating sirukumab and placebo, to preserve the blind).
  Interventions: Biological: sirukumab 50 mg; Drug: Placebo

INTERVENTIONS:
Biological: adalimumab 40 mg — SC injections
  Other Names: HUMIRA®
  Arms: Group 1 (adalimumab 40 mg)
Biological: sirukumab 100 mg — SC injections
  Other Names: CNTO 136
  Arms: Group 2 (sirukumab 100 mg)
Biological: sirukumab 50 mg — SC injections
  Other Names: CNTO 136
  Arms: Group 3 (sirukumab 50 mg)
Drug: Placebo — SC injections
  Arms: Group 2 (sirukumab 100 mg); Group 3 (sirukumab 50 mg)

SUMMARY:
The primary objective is to investigate the efficacy of sirukumab monotherapy compared with adalimumab monotherapy in biologic naïve subjects with active rheumatoid arthritis who are intolerant to methotrexate, who are considered inappropriate for treatment with methotrexate or who are inadequate responders to methotrexate.

DETAILED DESCRIPTION:
This is a randomized, double-blind, parallel-group, global, multicenter study of subcutaneous (SC) sirukumab monotherapy compared with adalimumab monotherapy in subjects with active rheumatoid arthritis. Approximately 510 subjects will be randomly assigned in a 1:1:1 ratio to receive treatment with adalimumab 40 mg SC every 2 weeks, sirukumab 100 mg SC every 2 weeks, or 50 mg SC every 4 weeks, with approximately 170 subjects per treatment group. At Week 16, subjects in all treatment groups who have < 20% improvement from baseline in both swollen and tender joint counts will qualify for early escape. The expected duration of the study is 68 weeks. This includes 52 weeks of treatment with study agent and 16 weeks of safety follow-up after the last study agent administration. The study will end when the last subject completes the last scheduled visit (Week 68 visit or completes the 16 week safety follow-up, whichever is later). Subject safety will be monitored through the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of rheumatoid arthritis (RA) for at least 6 months before screening
* Have moderately to severely active RA with at least 8 of 68 tender joints and 6 of 66 swollen joints, at screening and at baseline
* Have previous or current treatment with methotrexate (MTX) and are considered intolerant to MTX, and/or are considered inappropriate for treatment with MTX, (including MTX-naïve subjects for whom it is inappropriate to administer MTX) and/or an inadequate responder to methotrexate
* Must not have received MTX or any other non-biologic DMARD including but not limited to sulfasalazine, hydroxychloroquine, chloroquine, and bucillamine for at least 2 weeks prior to the first administration of the study agent
* C-reactive protein >= 10.00 mg/L or erythrocyte sedimentation rate >=28 mm/hr at screening

Exclusion Criteria:

* Has Functional Class IV as defined by the ACR Classification of Functional Status in Rheumatoid Arthritis
* Has ever received biologic therapy for RA, including but not limited to the following: TNF-alpha inhibitors, tocilizumab, rituximab, anakinra, abatacept
* Has ever used tofacitinib therapy or any other JAK inhibitor
* Has received intra-articular, intramuscular, or IV corticosteroids for RA, including adrenocorticotrophic hormone during the 4 weeks prior to first study agent administration
* Has received leflunomide within 24 months before the first study agent administration and has not undergone a drug elimination procedure, unless the M1 metabolite is measured and is undetectable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 559 (Actual)
Dates: Start 2014-04-04 (Actual); Primary Completion 2016-08-17 (Actual); Study Completion 2016-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (107):
- United States (42):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Arvin, California
  - El Cajon, California
  - Huntington Beach, California
  - Pleasanton, California
  - Thousand Oaks, California
  - Tustin, California
  - Whittier, California
  - Newark, Delaware
  - Aventura, Florida
  - Dunedin, Florida
  - Miami, Florida
  - New Port Richey, Florida
  - Palm Harbor, Florida
  - Plantation, Florida
  - Tampa, Florida
  - Kansas City, Kansas
  - Elizabethtown, Kentucky
  - Paducah, Kentucky
  - Frederick, Maryland
  - Wheaton, Maryland
  - St Louis, Missouri
  - Las Vegas, Nevada
  - Salisbury, North Carolina
  - Wilmington, North Carolina
  - Dayton, Ohio
  - Portland, Oregon
  - Duncansville, Pennsylvania
  - Wexford, Pennsylvania
  - Wyomissing, Pennsylvania
  - Jackson, Tennessee
  - Nashville, Tennessee
  - Austin, Texas
  - Carrollton, Texas
  - Corpus Christi, Texas
  - Cypress, Texas
  - Lubbock, Texas
  - McKinney, Texas
  - Mesquite, Texas
  - Chesapeake, Virginia
  - Clarksburg, West Virginia
- Bulgaria (2):
  - Rousse
  - Sofia
- Chile (2):
  - Port Montt
  - Temuco
- Colombia (3):
  - Barranquilla
  - Bogotá
  - Bucaramanga
- Germany (5):
  - Bad Doberan
  - Berlin
  - Cologne
  - Ratingen
  - Vogelsang-Gommern
- Hungary (2):
  - Debrecen
  - Gödöllő
- Lithuania (3):
  - Klaipėda
  - Šiauliai
  - Vilnius
- Mexico (4):
  - Chihuahua City
  - Guadalajara
  - Jalisco
  - Mexicali
- Chisinau, Moldova
- Poland (8):
  - Bydgoszcz
  - Bytom
  - Krakow
  - Lublin
  - Nadarzyn
  - Poznan
  - Warsaw
  - Wroclaw
- Romania (3):
  - Bucharest
  - Constanța
  - Ploieşti
- Russia (13):
  - Arkhangelsk
  - Kazan'
  - Kemerovo
  - Kursk
  - Moscow
  - Novosibirsk
  - Petrozavodsk
  - Ryazan
  - Saint Petersburg
  - Tomsk
  - Tver'
  - Vladimir
  - Yaroslavl
- Serbia (3):
  - Belgrade
  - Novi Sad
  - Zemun
- South Africa (4):
  - Cape Town
  - Durban
  - Kempton Park
  - Stellenbosch
- Spain (2):
  - A Coruña
  - Madrid
- Ukraine (10):
  - Chernihiv
  - Kryvyi Rih
  - Kyiv
  - Lviv
  - Odesa
  - Poltava
  - Sumy
  - Ternopil
  - Vinnytsia
  - Zaporizhzhia

REFERENCES:
- [Derived] Taylor PC, Schiff MH, Wang Q, Jiang Y, Zhuang Y, Kurrasch R, Daga S, Rao R, Tak PP, Hsu B. Efficacy and safety of monotherapy with sirukumab compared with adalimumab monotherapy in biologic-naive patients with active rheumatoid arthritis (SIRROUND-H): a randomised, double-blind, parallel-group, multinational, 52-week, phase 3 study. Ann Rheum Dis. 2018 May;77(5):658-666. doi: 10.1136/annrheumdis-2017-212496. Epub 2018 Feb 26. PMID 29483080

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 559 participants were randomized and treated. All participants received at least one administration of study treatment.
Groups:
- Adalimumab 40 mg: Participants received 40 milligram (mg) of adalimumab subcutaneously once every 2 weeks (q2w) for 52 weeks. Participants who met early escape (EE) criteria (had less than 20 percent improvement from baseline in swollen and tender joint counts) at Week 16 received adalimumab 40 mg once every week (q1w) through Week 52.
- Sirukumab 50 mg: Participants received 50 mg of sirukumab subcutaneously every 4 weeks (q4w) for 52 weeks and in between placebo SC injections was received at Weeks 2, 6, 10 and 14. Participants who met EE criteria at Week 16 received 100 mg sirukumab every 2 weeks (q2w) from Week 16 through Week 52 and placebo SC injections q2w between the sirukumab injections from Week 16 through Week 50.
- Sirukumab 100 mg: Participants received 100 mg of sirukumab subcutaneous injections at Weeks 0, 2, and every 2 weeks (q2w) through Week 52. Participants who met EE criteria at Week 16 received placebo injections q2w in between the sirukumab injections through Week 52.
Period: Overall Study
Arm/Group | Adalimumab 40 mg | Sirukumab 50 mg | Sirukumab 100 mg
Started | 186 | 186 | 187
Completed | 149 | 134 | 145
Not Completed | 37 | 52 | 42
Not completed — Adverse Event | 14 | 23 | 17
Not completed — Death | 0 | 1 | 1
Not completed — Lack of Efficacy | 7 | 4 | 4
Not completed — Lost to Follow-up | 0 | 2 | 1
Not completed — Physician Decision | 1 | 2 | 0
Not completed — Pregnancy | 1 | 2 | 2
Not completed — Withdrawal by Subject | 11 | 10 | 11
Not completed — Other | 3 | 8 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adalimumab 40 mg | Sirukumab 50 mg | Sirukumab 100 mg | Total
Number analyzed (Participants) | 186 | 186 | 187 | 559
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 163 | 159 | 164 | 486
  >=65 years | 23 | 27 | 23 | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.6 (12.15) | 52.5 (12.46) | 49.8 (12.31) | 51.6 (12.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 156 | 157 | 154 | 467
  Male | 30 | 29 | 33 | 92
Region of Enrollment [Number; unit: participants]
  Bulgaria | 1 | 1 | 0 | 2
  Chile | 5 | 2 | 3 | 10
  Colombia | 7 | 6 | 1 | 14
  Germany | 5 | 1 | 5 | 11
  Hungary | 0 | 1 | 2 | 3
  Lithuania | 12 | 15 | 9 | 36
  Mexico | 3 | 5 | 3 | 11
  Moldova | 2 | 6 | 4 | 12
  Poland | 21 | 17 | 20 | 58
  Romania | 4 | 5 | 4 | 13
  Russian Federation | 30 | 29 | 33 | 92
  Serbia | 20 | 19 | 26 | 65
  South Africa | 8 | 9 | 7 | 24
  Spain | 1 | 1 | 0 | 2
  Ukraine | 42 | 37 | 39 | 118
  United States | 25 | 32 | 31 | 88

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Disease Activity Index Score 28 (DAS28) Erythrocyte Sedimentation Rate (ESR) at Week 24
Description: The Disease Activity Index Score 28 using ESR [DAS28 (ESR)] is a derived score combining tender joints (28 joints), swollen joints (28 joints), ESR, and Patient's Global Assessment of Disease Activity. The 28 joints evaluated for swelling and tenderness were shoulder, elbow, wrist, MCP1, MCP2, MCP3, MCP4, MCP5, PIP1, PIP2, PIP3, PIP4, PIP5 joints of the upper right and upper left extremities as well as the knee joints of the lower right and lower left extremities. The DAS28-ESR is expressed on a score range of "0-10", with the minimum score= 0 (best) to maximum score= 10 (worst).
Time Frame: Baseline and Week 24
Population: Full analysis set was defined as all randomized participants who received at least 1 (partial or complete) dose of study agent. Participants with missing DAS28 (ESR) at baseline were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab 40 mg | Sirukumab 50 mg | Sirukumab 100 mg
Number analyzed (Participants) | 186 | 185 | 185
units on a scale
  Baseline | 6.89 (0.851) | 6.90 (0.881) | 6.91 (0.863)
  Change from Baseline at Week 24 | -2.19 (1.437) | -2.58 (1.524) | -2.96 (1.58)
Statistical Analysis 1: Comparison: Adalimumab 40 mg vs Sirukumab 100 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; LS mean difference = -0.76, 95% CI 2-sided [-1.07 to -0.46]
Statistical Analysis 2: Comparison: Adalimumab 40 mg vs Sirukumab 50 mg; Test type: Superiority or Other; p = 0.013, ANCOVA; Least Square (LS) mean difference = -0.39, 95% CI 2-sided [-0.69 to -0.08]

2. Primary Outcome: Percentage of Participants With an American College of Rheumatology (ACR) 50 Response at Week 24
Description: The ACR 50 Response is defined as greater than or equal to (>=) 50 percent (%) improvement in swollen joint count (66 joints) and tender joint count (68 joints) and >= 50% improvement in 3 of following 5 assessments: subject's assessment of pain using Visual Analog Scale (VAS) (0-10 millimeter [mm], 0 mm=no pain and 10 mm=worst possible pain), subject's global assessment of disease activity by using VAS (the scale ranges from 0 mm to 100 mm, [0 mm=no pain to 100 mm=worst possible pain]), physician's global assessment of disease activity using VAS (the scale ranges from 0 to 10, [0=no arthritis activity to 10=extremely active arthritis]), participant's assessment of physical function measured by Health Assessment Questionnaire-Disability Index (HAQ-DI) (the scale ranges from 0, indicating no difficulty, to 3, indicating inability to perform a task in that area) and serum C-Reactive Protein (CRP).
Time Frame: Week 24
Population: Full analysis set was defined as all randomized participants who received at least 1 (partial or complete) dose of study agent.
Measure: Number; unit: Percentage of participants
Arm/Group | Adalimumab 40 mg | Sirukumab 50 mg | Sirukumab 100 mg
Number analyzed (Participants) | 186 | 186 | 187
Percentage of participants | 31.7 | 26.9 | 35.3
Statistical Analysis 1: Comparison: Adalimumab 40 mg vs Sirukumab 50 mg; Test type: Superiority or Other; p = 0.306, Cochran-Mantel-Haenszel; Percentage Difference = -4.8, 95% CI 2-sided [-14.1 to 4.4]
Statistical Analysis 2: Comparison: Adalimumab 40 mg vs Sirukumab 100 mg; Test type: Superiority or Other; p = 0.464, Cochran-Mantel-Haenszel; Percentage Difference = 3.6, 95% CI 2-sided [-6 to 13.1]

3. Secondary Outcome: Percentage of Participants With Disease Activity Index Score 28 (DAS28) Using Erythrocyte Sedimentation Rate (ESR) Remission at Week 24
Description: The Disease Activity Index Score 28 using ESR [DAS28 (ESR)] is a derived score combining tender joints (28 joints), swollen joints (28 joints), ESR, and Patient's Global Assessment of Disease Activity. The 28 joints evaluated for swelling and tenderness were shoulder, elbow, wrist, MCP1, MCP2, MCP3, MCP4, MCP5, PIP1, PIP2, PIP3, PIP4, PIP5 joints of the upper right and upper left extremities as well as the knee joints of the lower right and lower left extremities. The DAS28-ESR is expressed on a score range of "0-10", with the minimum score= 0 (best) to maximum score= 10 (worst). The DAS28 (ESR) remission is defined as a DAS28 (ESR) value of less than 2.6 at a visit.
Time Frame: Week 24
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Adalimumab 40 mg | Sirukumab 50 mg | Sirukumab 100 mg
Number analyzed (Participants) | 186 | 186 | 187
Percentage of participants | 7.5 | 12.9 | 20.3
Statistical Analysis 1: Comparison: Adalimumab 40 mg vs Sirukumab 50 mg; Test type: Superiority or Other; p = 0.086, Cochran-Mantel-Haenszel; Percentage Difference = 5.4, 95% CI 2-sided [-0.7 to 11.4]
Statistical Analysis 2: Comparison: Adalimumab 40 mg vs Sirukumab 100 mg; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Percentage Difference = 12.8, 95% CI 2-sided [5.9 to 19.7]

4. Secondary Outcome: Percentage of Participants With an American College of Rheumatology (ACR) 20 Response at Week 24
Description: The ACR 20 Response is defined as >= 20% improvement in swollen joint count (66 joints) and tender joint count (68 joints) and >=20% improvement in 3 of following 5 assessments: subject's assessment of pain using VAS (0-10 mm, 0 mm=no pain and 10 mm=worst possible pain), subject's global assessment of disease activity by using VAS (the scale ranges from 0 mm to 100 mm, [0 mm=no pain to 100 mm=worst possible pain]), physician's global assessment of disease activity using VAS, subject's assessment of physical function measured by HAQ-DI, defined as a 20-question instrument assessing 8 functional areas. The derived HAQ-DI ranges from 0, indicating no difficulty, to 3, indicating inability to perform a task in that area) and serum CRP.
Time Frame: Week 24
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Adalimumab 40 mg | Sirukumab 50 mg | Sirukumab 100 mg
Number analyzed (Participants) | 186 | 186 | 187
Percentage of participants | 56.5 | 53.8 | 58.8
Statistical Analysis 1: Comparison: Adalimumab 40 mg vs Sirukumab 50 mg; Test type: Superiority or Other; p = 0.603, Cochran-Mantel-Haenszel; Percentage Difference = -2.7, 95% CI 2-sided [-12.8 to 7.4]
Statistical Analysis 2: Comparison: Adalimumab 40 mg vs Sirukumab 100 mg; Test type: Superiority or Other; p = 0.644, Cochran-Mantel-Haenszel; Percentage Difference = 2.4, 95% CI 2-sided [-7.6 to 12.3]

ADVERSE EVENTS:
Time Frame: Screening, up to Week 68
Description: Safety population included all participants who were randomized, received at least 1 (partial or complete) dose of double-blind study agent, and contributed any safety data after the start of study treatment.
Groups:
- Adalimumab 40 mg q2w Only: Participants received 40 mg of adalimumab subcutaneously q2w for 52 weeks.
- Adalimumab 40 mg q2w Then 40 mg q1w: Participants received 40 mg adalimumab subcutaneously q2w until Week 16 and received 40 mg adalimumab subcutaneously weekly (q1w) (due to EE) through Week 52.
- Sirukumab 50 mg q4w Only: Participants received 50 mg of sirukumab subcutaneously every four weeks (q4w) for 52 weeks.
- Sirukumab 50 mg q4w Then 100 mg q2w: Participants received 50 mg sirukumab until Week 16 and received 100 mg sirukumab subcutaneously q4w (due to EE or inadvertently) through Week 52.
Arm/Group | Adalimumab 40 mg q2w Only | Adalimumab 40 mg q2w Then 40 mg q1w | Adalimumab 40 mg | Sirukumab 50 mg q4w Only | Sirukumab 50 mg q4w Then 100 mg q2w | Sirukumab 50 mg | Sirukumab 100 mg
Serious Adverse Events (participants affected / at risk) | 15/173 | 1/13 | 16/186 | 23/160 | 6/26 | 29/186 | 22/187
Other Adverse Events (participants affected / at risk) | 71/173 | 3/13 | 74/186 | 79/160 | 13/26 | 92/186 | 86/187
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab 40 mg q2w Only (N=173) | Adalimumab 40 mg q2w Then 40 mg q1w (N=13) | Adalimumab 40 mg (N=186) | Sirukumab 50 mg q4w Only (N=160) | Sirukumab 50 mg q4w Then 100 mg q2w (N=26) | Sirukumab 50 mg (N=186) | Sirukumab 100 mg (N=187)
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 1 | 2 | 0 | 2 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Sinus node dysfunction (Cardiac disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diverticular perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Gastrointestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Subileus (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 2 | 0 | 2 | 0 | 0 | 0 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bursitis infective (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 2 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Erysipelas (Infections and infestations) | 1 | 0 | 1 | 0 | 1 | 1 | 0
Gastrointestinal bacterial infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Herpes ophthalmic (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Infectious pleural effusion (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 2 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 1 | 0 | 1 | 1
Pneumonia streptococcal (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 1 | 0 | 1 | 1 | 0 | 1 | 0
Pulpitis dental (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Tongue abscess (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Skin wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 0 | 1 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gliomatosis cerebri (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lacunar infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neuralgia (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Essential hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vasculitis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab 40 mg q2w Only (N=173) | Adalimumab 40 mg q2w Then 40 mg q1w (N=13) | Adalimumab 40 mg (N=186) | Sirukumab 50 mg q4w Only (N=160) | Sirukumab 50 mg q4w Then 100 mg q2w (N=26) | Sirukumab 50 mg (N=186) | Sirukumab 100 mg (N=187)
Neutropenia (Blood and lymphatic system disorders) | 4 | 0 | 4 | 16 | 1 | 17 | 11
Injection site erythema (General disorders) | 13 | 0 | 13 | 15 | 2 | 17 | 33
Injection site pruritus (General disorders) | 8 | 0 | 8 | 6 | 0 | 6 | 17
Injection site swelling (General disorders) | 4 | 0 | 4 | 3 | 1 | 4 | 11
Bronchitis (Infections and infestations) | 4 | 0 | 4 | 8 | 2 | 10 | 8
Nasopharyngitis (Infections and infestations) | 16 | 0 | 16 | 9 | 1 | 10 | 9
Upper respiratory tract infection (Infections and infestations) | 10 | 0 | 10 | 8 | 2 | 10 | 9
Alanine aminotransferase increased (Investigations) | 12 | 0 | 12 | 18 | 3 | 21 | 24
Aspartate aminotransferase increased (Investigations) | 11 | 0 | 11 | 9 | 4 | 13 | 20
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 17 | 0 | 17 | 17 | 3 | 20 | 15
Headache (Nervous system disorders) | 9 | 2 | 11 | 10 | 1 | 11 | 13
Hypertension (Vascular disorders) | 9 | 1 | 10 | 8 | 4 | 12 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.